CLINICAL TRIAL: NCT07390578
Title: Comparative Effect of Oxymetazoline 0.1% (Upneeq) and Brimonidine 0.025% (Lumify) on Upper Eyelid Position in Acquired Ptosis: A Randomized, Double-Masked, Crossover Study
Brief Title: Upneeq vs. Lumify Ptosis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00119513
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Acquired Ptosis
Keywords: Ptosis; Oxymetazoline; Brimonidine
MeSH Terms: conditions — Blepharoptosis | interventions — Oxymetazoline; Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Upneeq First, then Lumify (Experimental): Participants receive oxymetazoline 0.1% (Upneeq) at Visit 1 and brimonidine 0.025% (Lumify) at Visit 2.
  Interventions: Drug: Oxymetazoline 0.1% (Upneeq); Drug: Brimonidine 0.025% (Lumify)
- Lumify First, then Upneeq (Experimental): Participants receive brimonidine 0.025% (Lumify) at Visit 1 and oxymetazoline 0.1% (Upneeq) at Visit 2.
  Interventions: Drug: Oxymetazoline 0.1% (Upneeq); Drug: Brimonidine 0.025% (Lumify)

INTERVENTIONS:
Drug: Oxymetazoline 0.1% (Upneeq) — Single instillation of oxymetazoline 0.1% ophthalmic solution in both eyes.
Drug: Brimonidine 0.025% (Lumify) — Single instillation of brimonidine 0.025% ophthalmic solution in both eyes.

SUMMARY:
This study aims to compare the short-term effect of oxymetazoline 0.1% (Upneeq) versus brimonidine 0.025% (Lumify) on upper-eyelid position in adults with acquired ptosis. Participants will undergo standardized eyelid photography, receive a single dose of either Upneeq or Lumify in randomized order, and have repeat photographs approximately 60 minutes later. They will return for a second visit to receive the alternate medication using the same procedures. Eyelid height measurements will be obtained from coded images by masked graders. Data will be analyzed using paired statistical methods appropriate for a crossover design. Both medications are FDA-approved topical ophthalmic drops, and the study involves minimal risk with anticipated transient ocular irritation as the most common adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Adults age ≥18 years
* Acquired ptosis with MRD1 ≤ 2.5 mm in at least one eye
* Ability to complete both study visits (≥48 hours apart)
* Fluent in English
* Able to provide informed consent

Exclusion Criteria:

* Congenital ptosis or mechanical ptosis due to mass effect
* Ocular surgery within the past 6 months
* Significant active ocular surface disease
* Current contact lens wear on study days
* Known allergy to oxymetazoline or brimonidine
* Use of MAO inhibitors, α-blockers, or contraindicated medications
* Pregnancy or lactation
* Significant uncontrolled cardiovascular disease
* Any condition that may interfere with study procedures or data reliability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in upper-eyelid height (MRD1) (Upneeq vs. Lumify) | 60 minutes after instillation
  Change in MRD1 at ~60 minutes after drop instillation (Upneeq vs. Lumify)

SECONDARY OUTCOMES:
Change in palpebral fissure height (PFH) | 60 minutes after instillation
Number of participants with Conjunctival redness | 60 minutes after each medication
Participant-reported improvement in eyelid elevation or visual function | 60 minutes after each medication
  Participants will report eyelid elevation and visual function on a 0-10 numeric rating scale after each medication, where: 0 = no noticeable eyelid lift and 10 = maximal eyelid lift. For visual function: 0 = no improvement in vision and 10 = maximal improvement in vision.
Frequency of Adverse Events | 60 minutes after each medication
  Assess the safety and tolerability of a single dose of Upneeq and Lumify.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Dermarkarian, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No